CLINICAL TRIAL: NCT03768570
Title: A Randomized Phase II Trial Assessing Trimodality Therapy With or Without Adjuvant Durvalumab to Treat Patients With Muscle-Invasive Bladder Cancer
Brief Title: Trimodality Therapy With/Out Durvalumab to Treat Patients With Muscle-Invasive Bladder Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL13; 2019-001310-42 (EudraCT Number)
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-05

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surveillance (No Intervention)
- Durvalumab (Active Comparator)
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — 1500 mg IV on day 1 of 4 week cycle every 4 weeks for 12 months
  Arms: Durvalumab

SUMMARY:
The purpose of this study is to find out what effects durvalumab has on bladder cancer, combined with treatment after completion of surgery, chemotherapy and radiotherapy.

DETAILED DESCRIPTION:
This study is looking at whether a type of immunotherapy drug called durvalumab can be safely administered after initial treatment received by a patient. Durvalumab has been tested in many different types of cancers. Durvalumab works by allowing the immune system to detect cancer and reactivate the immune response. This may help to slow down the growth of cancer or may cause cancer cells to die. It is unclear if the addition of durvalumab is beneficial in patients with bladder cancer who have completed surgery, radiotherapy and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of urothelial carcinoma of the bladder. Patients with mixed histology (including small cell) and urothelial carcinoma are eligible. Patients with pure small cell carcinoma will be excluded.
* Stage T2-T4a N0M0 at time of diagnosis based on trans-urethral resection of bladder tumour, imaging, and/or bimanual examination under anesthesia.
* CT scan of the chest/abdomen/pelvis within 8 weeks from enrollment, showing no evidence of metastatic disease.
* Patients must be ≥ 18 years of age.
* Patients must have a life expectancy greater than 6 months.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 and a body weight of > 30kg.
* Patients must have adequate hematologic reserve: Platelet count ≥ 75 x 10^9/L, Absolute neutrophils ≥ 1.0 x 10^9/L. Anemia will be corrected to minimum hemoglobin of 90 g/L with red cell transfusions, if necessary.
* Patients must have an estimated creatinine clearance (Cockcroft-Gault Equation) ≥ 30 ml/min.
* Patients must have adequate liver function with a bilirubin ≤ 1.5 ULN (if confirmed Gilbert's, eligible providing bilirubin ≤ 3 x UNL) and AST/ALT (SGOT/SGPT) < 2.5 x the upper normal limit.
* All patients must have a tumour block from their primary tumour available and consent to release the block/cores/cut slides for correlative analyses ( and the centre/pathologist must have agreed to the submission of the specimen(s).
* Patients have completed prior trimodality therapy (TMT) consisting of surgery, chemotherapy and radiation therapy treatment prior to enrollment. Patient should start treatment within 42 days after completion of TMT.
* Patients must have undergone a transurethral resection prior to study enrollment.
* Patient may have completed up to 4 cycles of cisplatin-based neo-adjuvant chemotherapy. Adjuvant chemotherapy is not permitted. Patients will have received cisplatin, given intravenously during the radiation therapy. OR Patients may have received fluorouracil and mitomycin given intravenously once weekly or gemcitabine as an alternative to cisplatin during radiotherapy.
* The following are radiotherapy guidelines for patients treated on study. Patients will be treated to radical treatment doses using IMRT, VMAT or 4 field conformal techniques. Planning will be based on CT planning. IGRT is recommended during the radiotherapy treatment. Recognizing differences in usual radiotherapy doses used in the various participating countries and centres the following would be acceptable doses in this study. The bladder CTV will include the whole empty bladder and any extravesical extension. PTV expansion will be a minimum of 0.75 cm right, left and inferiorly, 1.5 cm Anteriorly and superiorly and 1 cm posteriorly. These minimum expansions are with Cone beam verification. For patients undergoing RT without image-guided verification 1.5 cm expansion in all directions is recommended. Acceptable doses for this study include:

  * Bladder only: 64-66 Gy in 32-33 fractions over 6.5 weeks; 50-55 Gy in 20 fractions over 4 weeks
  * Pelvis and bladder: 45-46 Gy to pelvic nodes + 17-20 Gy bladder boost in 33-35 fractions over 6.5-7 wks [Note: minimal nodal dose (if used) is 44 Gy in 32f or 40 Gy in 20f]
* Patients receiving concurrent bladder boost: pelvis dose 40 Gy and bladder dose 50 Gy given in 20 fractions over 4 weeks. Adaptive radiotherapy techniques would be acceptable.
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires in either English, French or Spanish.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits placed on patients being considered for this trial.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient enrollment.
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method during and for 3 months following treatment.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

* Pre-existing medical conditions precluding treatment.
* Pregnancy or lactating mothers.
* Received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-PD-L1, including durvalumab anti-programmed cell death-ligand 2 (anti-PD-L2), anti-CD137 (4-1BB ligand, a member of the Tumour Necrosis Factor Receptor [TNFR] family), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease (e.g. colitis or Crohn's disease: not due to radiation reaction), diverticulitis with the exception of diverticulosis, celiac disease (controlled by diet alone) or other serious gastrointestinal chronic conditions associated with diarrhea), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis), rheumatoid arthritis, hypophysitis, uveitis, etc., within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

  * Patients with alopecia;
  * Patients with Grave's disease, vitiligo or psoriasis not requiring systemic treatment (within the last 2 years);
  * Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement;
  * Any chronic skin condition that does not require systemic therapy.
* Patients with active or uncontrolled intercurrent illness including, but not limited to:

  * cardiac dysfunction (symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia);
  * active peptic ulcer disease or gastritis;
  * active bleeding diatheses;
  * psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent;
  * known history of previous clinical diagnosis of tuberculosis;
  * known active human immunodeficiency virus infection (positive HIV 1/2 antibodies). HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible;
  * known active hepatitis B infection (positive HBV surface antigen (HBsAg). Patients with a past or resolved HBV infection (defined as presence of hepatitis B core antibody (anti-HBc) and absence of HBsAg) are eligible;
  * known active hepatitis C infection. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* History of primary immunodeficiency, history of allogenic organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 28 days of randomization or a prior history of severe (grade 3 or 4) immune mediated toxicity from other immune therapy or grade ≥ 3 infusion reaction.
* Current or prior use of immunosuppressive medication within 28 days of study entry, with the exceptions of intranasal and inhaled corticosteroids or systemic chronic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Corticosteroids used on study for anti-emetic purpose are allowed. Corticosteroids as premedication for hypersensitivity reactions (e.g. computed tomography [CT] scan premedication) are allowed.
* Peripheral neuropathy ≥ grade 2 (CTCAE v5.0).
* History of allergic or hypersensitivity reactions to any study drug or their excipients.
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 470 msec in screening ECG measured using standard institutional method or history of familial long QT syndrome.
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline CT scan.
* Any active disease condition which would render the protocol treatment dangerous or impair the ability of the patient to receive protocol therapy.
* Any condition (e.g. psychological, geographical, etc.) that does not permit compliance with the protocol.
* Live attenuated vaccination administered within 30 days prior to randomization.
* Any prior carboplatin based therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 5 years
  defined as the time from the randomization to the time of the first event that is either recurrent (local or distant) bladder cancer, a new primary bladder cancer or death from any cause

SECONDARY OUTCOMES:
Non-muscle invasive bladder cancer recurrence rate | 5 years
Loco-regional control rate between study arms at the 12 week visit | 5 years
  defined as proportion of patients with a confirmed locoregional complete response at 3 months post randomization
Patterns of disease recurrence between study arms | 5 years
  The two treatment arms will be compared using the log-rank test stratified by ECOG Performance Status (0, 1 vs. 2+), Neoadjuvant chemotherapy (Yes/No), whole bladder versus partial bladder versus bladder plus regional lymph nodes RT field, and disease stage (T2 vs T3/4). A table will be presented summarizing the patterns of disease recurrence by treatment arms
Compare overall and bladder intact disease-free survival between study arms | 5 years
Metastasis-free survival between study arms | 5 years
Number and severity of adverse events between study arms | 5 years
Quality of Life between treatment arms using Functional Assessment of Cancer Therapy-Bladder Cancer (FACT-BL) questionnaire | 5 years
  It consists of 39 questions, of which 12 are specific to bladder cancer. The questionnaire consists of 5 subscales: physical well-being (PWB), social/family well-being (SWB), emotional well-being (EWB), functional well-being (FWB), and a final subscale focusing specifically on bladder cancer.
Cost-effectiveness between study arms | 5 years
  Estimate an incremental cost-effectiveness ratio reported as a difference in cost per Disease free survival-year gained of durvalumab vs. surveillance. analyses will focus on the incremental cost-effectiveness of durvalumab from a government payer perspective, over a disease-free survival time horizon by prospectively collecting economic and resource utilization information during the clinical trial.
Cost-utility between study arms | 5 years
  A partitioned-survival model (Markov model) will be developed using data obtained from the trial. Different parametric models will be evaluated to fit data from the trial in order to evaluate the incremental cost-utility over a 3-, 5- and 10-y horizon.

CONTACTS AND LOCATIONS:
Overall Officials: Wassim Kassouf, Study Chair — The Research Institute of the McGill University, Montreal QC Canada
Locations (31):
- Canada (15):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre/, Thunder Bay, Ontario
  - University Health Network, Toronto, Ontario
  - The Jewish General Hospital, Montreal, Quebec
  - The Research Institute of the McGill University, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Spain (8):
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - Instituto Valenciano de Oncologia, Valencia
- United Kingdom (8):
  - Royal Devon and Exeter Hospital, Exeter, Devon
  - Royal Cornwall Hospitals NHS Trust, Cornwall, England
  - Royal Preston Hospital, Lancashire, England
  - Charing Cross Hospital, London, England
  - The Christie NHS Foundation Trust, Manchester, England
  - The Royal Marsden NHS Foundation Trust - Sutton, Surrey, England
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Nottingham University Hospitals City Hospital Campus, Nottingham

IPD SHARING:
Plan to Share IPD: No